CLINICAL TRIAL: NCT03728998
Title: Can Non-invasive Measurement of Cardiac Index, Stroke Volume and Systemic Vascular Resistance Contribute to Better Tailoring of Treatment in Patients Presenting With Sepsis to the ED?
Brief Title: Non-invasive Measurement of CO in Patients With Uncomplicated Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: nWMO271
Record Dates: First submitted 2018-07-17; First posted 2018-11-02 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2018-06

CONDITIONS: Sepsis
Keywords: Passive leg raise; Fluid responsiveness; Cardiac output, non-invasive; Emergency Department
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLR & Clearsight measurements (Other): All patients 16years or older presenting to the ED with uncomplicated sepsis (see inclusion and exclusion criteria) will undergo a Passive Leg Raise (PLR, non-invasive) and multiple measurements by the Clearsight non-invasive hemodynamic monitoring system. Followed by a fluid challenge (common practice; non interventional)
  Interventions: Other: Passive leg raise (PLR); Other: Clearsight non-invasive hemodynamic monitoring system

INTERVENTIONS:
Other: Passive leg raise (PLR) — A PLR will simulate an autotransfusion of 250-300 cc.
  * 1. Starting in semi-succumbed position (45 degree head-up)
  * 2. PLR is performed by lowering head-end and putting a for this purpose designed device of 45 degrees under the patients legs. The PLR is non-invasive.
Other: Clearsight non-invasive hemodynamic monitoring system — 3 baseline readings will be done for CO, CI, SV and SVR, separated by one minute intervals. Subsequently, the standardized passive leg-raise test will be performed and measurements of CO, CI, SV and SVR will be repeated at 30, 60, 90 and 120 seconds. Then the patient is repositioned to his original position, and after two minutes another reading of CO, CI, SV and SVR is done. Then all patients will receive a fluid challenge of 500cc natriumchloride 0.9% IV, considered as normal treatment/ common practice in our ED. 120 seconds after finishing the fluid challenge the final reading of CO, CI, SV and SVR is done.

SUMMARY:
Little is known about the optimal fluid therapy of patients with uncomplicated sepsis. Most recommendations are extrapolated from studies performed in patients with septic shock. Therefore, it is unknown how effective our current fluid therapy is. Furthermore, current therapy is not tailored to individual needs. The aim of the current study is to investigate the added value of non-invasive measurements of (dynamic) circulatory parameters in the treatment of a convenience sample of sepsis patients presenting to the ED.

ELIGIBILITY:
Inclusion Criteria:

At presentation in the ED:

* there has to be evidence of an infection: -temp <36 or >38 without an obvious cause for hypo-or hyperthermia
* There has to be evidence of organ dysfunction by the presence of at least one of the following criteria: altered mental state, hypoxia (spo2<94% or 5% lower than baseline), lactate >2 mmol/l in ABGA or VBGA directly drawn after presentation, hypotension (MAP<65 mmHg or SBP<100mmHg), or a respiratory rate>22/min.

Exclusion Criteria:

* Age<16
* Patients with septic shock (i.e. who remained hypotensive after fluid bolus administration, needing vasopressor therapy to obtain a MAP>65 in the presence of a lactate >2. (i.e. septic shock) These will be excluded afterwards, but will be shown in an inclusion flowchart.
* Subjects for whom it is impossible to obtain a reliable signal for Clearsight measurements.
* Increased abdominal pressures
* Need for immediate ventilatory support or surgery
* Presence of an acute cerebral event, acute coronary syndrome, acute pulmonary edema, status asthmaticus, active gastrointestinal bleed, trauma
* Known metastatic cancer
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects in whom a passive leg raise test resulted in a 15% or more improvement in cardiac index measured by the Clearsight non-invasive hemodynamic monitoring system. | 1 hour
  3 baseline readings will be done for CI separated by one minute intervals. Subsequently, the standardized passive leg-raise test will be performed and measurements of CI will be repeated at 30, 60, 90 and 120 seconds. Then the patient is repositioned to his original position, and after two minutes another reading of CI is done. A difference of 15% or more is found to be clinically significant.

SECONDARY OUTCOMES:
The ability of non-invasively measured baseline CO, CI, SVR and SV to predict fluid-responsiveness correctly (measurements by the Clearsight non-invasive hemodynamic monitoring system). | 1 hour
  3 baseline readings will be done for CO, CI, SV and SVR, separated by one minute intervals. Subsequently, the standardized passive leg-raise test will be performed and measurements of CO, CI, SV and SVR will be repeated at 30, 60, 90 and 120 seconds. Then the patient is repositioned to his original position, and after two minutes another reading of CO, CI, SV and SVR is done. Then all patients will receive a fluid challenge of 500cc natriumchloride 0.9% IV, considered as normal treatment/ common practice in our ED. 120 seconds after finishing the fluid challenge the final reading of CO, CI, SV and SVR is done.

CONTACTS AND LOCATIONS:
Overall Officials: Ewoud ter Avest, MD, PhD, Principal Investigator — Medisch Centrum Leeuwarden
Locations (1):
- Medisch Centrum Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided